CLINICAL TRIAL: NCT02456558
Title: A Phase Ib Randomized, Double-blind, Placebo-controlled, Ascending Sequential Dose, Adaptive Design Study to Evaluate the Safety, Antiretroviral Activity, and Pharmacokinetics of Intravenous Deferiprone in Treatment-Naïve HIV-Positive Subjects
Brief Title: Evaluation of the Safety, Efficacy, and Pharmacokinetics of Intravenous Deferiprone in HIV-Positive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LA44-0114
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Asymptomatic HIV Infection
Keywords: HIV infection; antiretroviral drugs; deferiprone; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Isoflurophate; Deferiprone; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous deferiprone, 1.5 g (Experimental): Subjects in this arm will receive an infusion of intravenous deferiprone at a dose of 1.5 g, twice-daily
  Interventions: Drug: Intravenous deferiprone
- Intravenous deferiprone, 2 g (Experimental): Subjects in this arm will receive an infusion of intravenous deferiprone at a dose of 2 g, twice-daily
  Interventions: Drug: Intravenous deferiprone
- Placebo (Placebo Comparator): Subjects in this arm will receive an infusion of placebo twice-daily for 10 days, at a volume equivalent to that of the active product in the respective cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous deferiprone — In Cohort 1, the subjects who were randomized to get active product will receive deferiprone at a dose of 1.5 g per infusion, and if there are no significant safety concerns, the subjects in Cohort 2 who were randomized to get active product will receive it a a dose of 2 g per infusion.
  Other Names: IV DFP; Deferiprone injection, solution
  Arms: Intravenous deferiprone, 1.5 g; Intravenous deferiprone, 2 g
Drug: Placebo — In both cohorts, the subjects who were randomized to get placebo will receive an infusion of placebo solution that is equal in volume to that of the active product.
  Other Names: Normal saline solution (0.9% w/v NaCl)
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, antiretroviral activity, pharmacokinetics, and pharmacodynamics of an intravenous formulation of deferiprone in HIV-infected subjects.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized trial in 30 asymptomatic HIV-positive adults. There are two sequential cohorts, in which subjects will receive either one of 2 doses of deferiprone or placebo twice daily.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* HIV treatment-naïve: no previous treatment with a combination anti-retroviral therapy (cART) or highly active anti-retroviral therapy (HAART) regimen
* HIV-1 RNA > 10,000 copies/mL
* ALT or AST ≤ 2.0 x upper limit of normal range, and bilirubin within normal range
* Body mass index (BMI) of 18.5 to 30.0 kg/m^2
* Absolute neutrophil count at baseline of ≥1.0 x 10^9/L (black African population only) or ≥1.5 x 10^9/L (all other races)

Exclusion Criteria:

* Evidence of AIDS-associated illness, excluding superficial candidiasis
* CD4+ T-cell count of < 350/mm^3
* Positive for active or latent tuberculosis, as determined by the QuantiFERON®-TB Gold test
* Active, serious infections (other than HIV-1 infection) within the 30 days prior to screening
* Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis virus C (HCV) antibodies
* History or presence of malignancy
* A serious, unstable chronic illness during the past 3 months before screening
* A serious, unresolved acute illness at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV viral load | Day 1 to Day 56
Change from baseline in CD4+ T-cell count | Day 1 to Day 56
Change from baseline in level of HIV DNA in peripheral blood mononucleated cells | Day 1 to Day 56
Proportion of subjects withdrawn due to the need for rescue medication | Day 1 to Day 56
Number of subjects with adverse events | Day 1 to Day 56

SECONDARY OUTCOMES:
The pharmacokinetics parameters of Cmax, Tmax, and AUC0-∞, and T1/2 for deferiprone will be determined pre-dose and at specified time points post-dose | 10-hour interval

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - VxPharma, Pretoria